CLINICAL TRIAL: NCT02491190
Title: Using Multimedia Digital Health to Enable and Engage Pediatric Inpatients and Their Parents: A Pilot Study
Brief Title: Using Multimedia Digital Health to Enable and Engage Pediatric Inpatients and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-16151
Record Dates: First submitted 2015-06-26; First posted 2015-07-07 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Inpatient Pediatric Engagement and Shared Decision-Making

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Empower educational module: After the patient activation measure/s are collected, for parents or patients assigned to the intervention arm, they will be given an opportunity to launch the EMPOWER video and interactive powerpoint. They will be able to pause on reviewing the educational material and come back to it, as with other assigned education, and they will be able to review it again if they would like. Discharge surveys will be assigned 24 hours prior to the estimated discharge time in Apex. Oneview will display notifications that the surveys have been assigned.
  Interventions: Behavioral: EMPOWER Educational Module
- Control (No Intervention): Standard care: Those who opt to participate in the study will be randomly assigned to receive standard features of the media center (control group), or standard features plus the educational module intervention. They will complete online (1) a baseline patient activation survey (for patients old enough to complete and for caregivers) at the start of their participation, and (2) an end-of-study survey pre-discharge or at the end of the study period.

INTERVENTIONS:
Behavioral: EMPOWER Educational Module — Evidence-based video module delivering content of the Right Question intervention from Deen et al. (2011)
  Arms: Treatment

SUMMARY:
This project leverages digital health technology to support patient engagement and shared decision-making between families, patients, and providers. The investigators will start by finalizing the educational module and adding randomization for the trial (Aim 1). The investigators will then complete iterative user testing in the live system through measurement of educational module views and usability feedback interviews with 20 end users (Aim 2). The investigators will then conduct a randomized controlled trial to test the impact of the educational module on existing measures of patient engagement (Aim 3). The hypothesis is that parents who receive the educational module will have higher scores on shared decision-making, patient activation and overall patient experience.

DETAILED DESCRIPTION:
Hospitals are not consistently patient centered, contributing to worse outcomes and a sense of loss of control. Prior interventions that promote patient-centered care focused on provider and hospital factors vs. engaging patients directly. No project to date has capitalized on digital health technology to engage families in shared decision-making and patient engagement. The goal of the proposed randomized controlled trial is to test the impact of an evidence-based educational module delivered using an interactive patient-facing IT platform, on measures of patient engagement and shared decision-making. The platform was developed for the UCSF Benioff Children's Hospital by OneView, Inc. and includes an educational module that promotes shared decision-making through orientation to the hospital and evidence-based teaching on engaging with providers. This study will provide pilot data for a large-scale trial measuring the impact of the system on patient engagement. The investigators will start by finalizing the educational module and adding randomization for the trial (Aim 1). The investigators will then complete iterative user testing in the live system through measurement of educational module views and usability feedback interviews with 20 end users (Aim 2). The investigators will then conduct a randomized controlled trial to test the impact of the educational module on existing measures of patient engagement (Aim 3). Our hypothesis is that parents who receive the educational module will have higher scores on shared decision-making, patient activation and overall patient experience. The eligible study population is all pediatric and newborn inpatients and their caregivers from June 2015 - August 2015. The investigators anticipate needing a sample size of 100, 50 in each arm. This pilot will generate key information on the platform's feasibility and acceptability and initial data on effect sizes to power future large-scale grants.

ELIGIBILITY:
Inclusion Criteria:

* An admitted patient (up to age 22) or caregiver (up to 95) of an admitted patient at Benioff Children's Hospital in the acute care units, the pediatric hematology-oncology units, or the transitional care units, admitted to the hospital within the past 72 hours.

Exclusion Criteria:

* Was already admitted and discharged during the study period.
* Not an English speaker.
* Not having a parent or legal guardian present or available by phone to give consent for those <18 years of age.
* Patient is in foster care.

Max Age: 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in activation as measured with the Parent Patient Activation Measure (PPAM) | Measured at enrollment, and at hospital discharge--duration of hospital stay is an average of 3 days. Calculated as change in PPAM scores.

SECONDARY OUTCOMES:
Quality of Shared Decision-Making measured using the CollaboRATE 3-item scale | Measured at discharge, an average of 3 days after study enrollment
Quality of Shared Decision-Making measured using M-PICS scores | Measured at discharge, an average of 3 days after study enrollment
Length of Stay obtained from the Epic electronic health record | Measured at discharge, an average of 3 days after study enrollment
30-day readmission obtained from the Epic electronic health record | Measured 30 days after discharge. Discharge occurs an average of 3 days after study enrollment
  This is a binary measure assessing whether the patient was readmitted to the hospital (Benioff Children' Hospital) within 30 days after discharge date.
Study Recruitment Rate | Baseline
  Number of patients with at least one person agreeing to participate (either a family member or a child) / Number of eligible patients who were assigned the study introduction materials in the hospital electronic educational center
Study Retention | Measured at discharge, an average of 3 days after study enrollment
  Number of participants who complete the survey capturing the second patient activation measure prior to hospital discharge / Number of participants who completed the first Patient Activation Measure
Engagement with the Educational Module | Duration of the hospital stay, an average of 3 days
  Number of participants viewing the EMPOWER educational module (intervention) at least once / Number of patients assigned the module. Data from the OneView system
Repeated Engagement with the Education Module | Duration of the hospital stay, an average of 3 days
  Number of views of the educational module for participants who viewed it at least once

CONTACTS AND LOCATIONS:
Overall Officials: Naomi S. Bardach, MD, MAS, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pennarola BW, Rodday AM, Mayer DK, Ratichek SJ, Davies SM, Syrjala KL, Patel S, Bingen K, Kupst MJ, Schwartz L, Guinan EC, Hibbard JH, Parsons SK; HSCT-CHESS Study. Factors associated with parental activation in pediatric hematopoietic stem cell transplant. Med Care Res Rev. 2012 Apr;69(2):194-214. doi: 10.1177/1077558711431460. Epub 2011 Dec 26. PMID 22203645
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Alegria M, Polo A, Gao S, Santana L, Rothstein D, Jimenez A, Hunter ML, Mendieta F, Oddo V, Normand SL. Evaluation of a patient activation and empowerment intervention in mental health care. Med Care. 2008 Mar;46(3):247-56. doi: 10.1097/MLR.0b013e318158af52. PMID 18388839
- [Background] Deen D, Lu WH, Rothstein D, Santana L, Gold MR. Asking questions: the effect of a brief intervention in community health centers on patient activation. Patient Educ Couns. 2011 Aug;84(2):257-60. doi: 10.1016/j.pec.2010.07.026. Epub 2010 Aug 25. PMID 20800414
- [Background] Smith MY, Winkel G, Egert J, Diaz-Wionczek M, DuHamel KN. Patient-physician communication in the context of persistent pain: validation of a modified version of the patients' Perceived Involvement in Care Scale. J Pain Symptom Manage. 2006 Jul;32(1):71-81. doi: 10.1016/j.jpainsymman.2006.01.007. PMID 16824987
- [Background] Alegria M, Sribney W, Perez D, Laderman M, Keefe K. The role of patient activation on patient-provider communication and quality of care for US and foreign born Latino patients. J Gen Intern Med. 2009 Nov;24 Suppl 3(Suppl 3):534-41. doi: 10.1007/s11606-009-1074-x. PMID 19842003
- [Background] Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. Health Serv Res. 2005 Dec;40(6 Pt 1):1918-30. doi: 10.1111/j.1475-6773.2005.00438.x. PMID 16336556
- [Background] Barr PJ, Thompson R, Walsh T, Grande SW, Ozanne EM, Elwyn G. The psychometric properties of CollaboRATE: a fast and frugal patient-reported measure of the shared decision-making process. J Med Internet Res. 2014 Jan 3;16(1):e2. doi: 10.2196/jmir.3085. PMID 24389354
- [Derived] Bardach NS, Lam R, Jasik CB. Assessment of automated clinical trial recruitment and enrolment using patient-facing technology. BMJ Health Care Inform. 2021 Jan;28(1):e100076. doi: 10.1136/bmjhci-2019-100076. PMID 33504589